CLINICAL TRIAL: NCT05223088
Title: Tislelizumab Combined With Apatinib and Oxaliplatin Plus S1 as Neoadjuvant Therapy for Borrmann IV、Large Borrmann III Type and Bulky N Positive Advanced Gastric Cancer: a Single-arm, Prospective, Multicenter Trial (TAOS-3B-Trial)
Brief Title: Tislelizumab Combined With Apatinib and Oxaliplatin Plus S1 as Neoadjuvant Therapy for Borrmann IV、Large Borrmann III Type and Bulky N Positive Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAOS-3B
Record Dates: First submitted 2022-01-23; First posted 2022-02-03 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Immunotherapy; Gastrict Cancer
MeSH Terms: interventions — tislelizumab; apatinib; Oxaliplatin; Tegafur

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with apatinib and oxaliplatin plus S1 (Experimental): Neoadjuvant immunotherapy, PD-1, plus apatinib and oxaliplatin plus S1 will be applied to patients with Borrmann IV、large Borrmann III type and Bulky N positive advanced gastric cancer before surgery.
  Interventions: Drug: Tislelizumab; Drug: Apatinib Mesylate; Drug: oxaliplatin; Drug: Tegafur

INTERVENTIONS:
Drug: Tislelizumab — Participants will receive Tislelizumab, 200mg, intravenously over 30 - 60 minutes, day 1 of every 3 weeks for 3-6 weeks. Discontinuation will be considered due to toxicity, withdrawal of consent, or end of study. Every 3-week treatment period was considered to be a cycle.
Drug: Apatinib Mesylate — Participants will receive apatinib, 250mg, qd，every 3 weeks for 2-5 weeks.
Drug: oxaliplatin — Participants will receive oxaliplatin, 130mg/m2, day 1 of every 3 weeks for 3-6 weeks.
Drug: Tegafur — Participants will receive Tegafur, day 1-14 of every 3 weeks for 3-6 weeks.

SUMMARY:
To evaluate the clinical efficacy and safety of Tislelizumab combined with apatinib mesylate, oxaliplatin plus S1.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years of age
* Histologically confirmed gastric adenocarcinoma was diagnosed in patients with locally advanced gastric cancer with tumor volume >5cm Borrmann III, Borrmann IV and BulkyN according to AJCC Version 8
* measurable lesions at least should be detected by CT/MRI examination in accordance with the RECIST1.1.
* ECOG（Eastern Cooperative Oncology Group）PS（Performance Status）:0-1 scores;
* No previous surgical treatment, anti-tumor chemoradiotherapy/immunotherapy was performed
* Preoperative endoscopic examination confirmed no positive peritoneal implantation metastasis and exfoliated cells
* the expected survival time is more than 6 months
* the main organ function is normal, which should meet the following criteria:

  1. HB≥ 9g/dL
  2. ANC≥1.5×109/L
  3. PLT≥100×109/L
  4. TBIL≤1.5 normal upper limit ULN ；or TBIL>ULN but BIL≤ULN
  5. ALT and AST≤2.5 ULN（ALT or AST ≤5×ULN was allowed in patients with liver metastasis）
  6. Cr≤1.5 ULN，CCR（creatinine clearance rate）≥60ml/min(Cockcroft-Gault formula)
  7. Good coagulation function, defined as international standardized ratio (INR) or prothrombin time (PT) ≤1.5 ULN
  8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range.If the baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range may be enrolled;
  9. The myocardial enzyme profile is within the normal range (if the investigator comprehensively determines that the simple laboratory abnormality is not clinically significant, it is allowed to be included in the group
* For women of reproductive age, a urine or serum pregnancy test with negative results should be performed within 3 days prior to receiving the first study drug administration (day 1 of cycle 1).If a urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is requested.Women of childbearing age were defined as at least 1 year after menopause or having undergone surgical sterilization or hysterectomy;。
* If there is a risk of conception, all subjects (both men and women) are required to use a contraceptive with an annual failure rate of less than 1% throughout the treatment period up to 120 days after the last study drug (or 180 days after the last chemotherapeutic drug)
* participants is willing to participate in this study, sign the informed consent, have good compliance, cooperate with follow-up.

Exclusion Criteria:

* Diagnosis of malignant diseases other than gastric cancer within 5 years prior to first administration (excluding radical basal cell carcinoma of the skin, squamous carcinoma of the skin, and/or radical resectable carcinoma in situ);
* Significant clinical bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer or vasculitis, etc. occurred within 3 months before enrollment. If fecal occult blood was positive at baseline, reexamination could be performed; if it was still positive after reexamination, gastroscopy was required
* Prior treatment: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs that target another stimulating or co-inhibiting T-cell receptor (e.g., CTLA-4, OX-40, CD137);
* A history of immunodeficiency, including HIV testing positive.
* Is currently participating in an interventional clinical study or has been treated with another study drug or study device in the 4 weeks prior to initial dosing.
* Patients who had a history of cardiovascular and cerebrovascular diseases and were still taking thrombolytic drugs or anticoagulants orally.
* HER2 positive is known;
* Patients with previous gastrointestinal perforation, abdominal abscess or recent intestinal obstruction (within 3 months) or imaging or clinical symptoms suggesting intestinal obstruction;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Total/moderate tumor regression rate under pathology | 4 weeks after surgery
  Primary tumor or lymph node surgery specimen pathological examination without residual tumor cell

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At the end of Cycle 3 (each cycle is 21 days)
  Objective Response Rate Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor
Overall survival (OS) | every 3 months (up to 24 months) ]
  Defined from date of Signing ICF to date of first documentation of death from any cause or censored at the date of the last follow-up.
  Defined from date of Signing ICF to date of first documentation of death from any cause or censored at the date of the last follow-up.
  Defined from date of Signing ICF to date of first documentation of death from any cause or censored at the date of the last follow-up.
  Defined from date of Signing ICF to date of first documentation of death from any cause or censored at the date of the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian cancer hospital, Fuzhou, China